CLINICAL TRIAL: NCT00532246
Title: A Study of Carotid Artery Intima-Media Thickness Following Exposure to Raloxifene HCl or Placebo
Brief Title: Carotid Artery Intima-Media Thickness Following Exposure to Raloxifene or Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8135; H3S-MC-GGLE
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Osteoporosis, Post-Menopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): raloxifene
  Interventions: Drug: raloxifene
- B (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: raloxifene
  Other Names: LY139481
  Arms: A
Drug: Placebo
  Arms: B

SUMMARY:
The purpose of this study is to measure carotid artery IMT at a single visit in a subset of women previously enrolled in the CORE (H3S-MC-GGJY) trial

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed the Eli Lilly and Company clinical trial CORE (H3S-MC-GGJY) inclusive of visit 5, in one of the 9 participating study sites in California.
* Patients must have been dispensed study drug in the CORE trial (H3S-MC-GGJY).

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Have previously withdrawn from this exploratory study or any other study investigating raloxifene
* Are employed by Eli Lilly and Company (that is, employees, temporary contract workers, or designees responsible for the conduct the study). Immediate family of Eli Lilly and Company employees may participate in Lilly-sponsored clinical trials, but are not permitted to participate at an Eli Lilly and Company facility. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Are investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2003-03; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that in postmenopausal women with osteoporosis who took lipid lowering meds for more than 6 months > 80% compliant with study drug during CORE trial, mean carotid IMT will be lower in patients treated with raloxifene than placebo

SECONDARY OUTCOMES:
To test the hypothesis that, in postmenopausal women with osteoporosis, mean carotid IMT will be significantly lower in patients treated with raloxifene as compared to mean carotid IMT in patients treated with placebo in the following:
All enrolled patients who have not been exposed to lipid lowering medication for more than 6 months while in the CORE trial, regardless of study drug compliance.
All enrolled patients, regardless of lipid lowering drug exposure or compliance with study drug while in CORE
All enrolled patients who were at least 80% compliant with study drug while in CORE, regardless of use of lipid lowering therapy

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Menlo Park, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Walnut Creek, California

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com